CLINICAL TRIAL: NCT02128347
Title: Effectiveness of an Online Portal for Delivery of Care to Home Dialysis Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Karthik Tennankore (Other)
Responsible Party: Sponsor-Investigator, Karthik Tennankore, Assistant Professor, Division of Nephrology, Department of Medicine, Nova Scotia Health Authority
Organization: Nova Scotia Health Authority (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: eportal 2014-316
Record Dates: First submitted 2014-04-29; First posted 2014-05-01 (Estimated); Last update posted 2016-07-26 (Estimated); Status verified 2016-07

CONDITIONS: Hemodialysis, Home; Peritoneal Dialysis
Keywords: Hemodialysis, Home; Peritoneal Dialysis; Telemedicine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Electronic Patient Portal (Other): RelayHealth is a web-based application that allows patients and healthcare workers to communicate through a secure, password protected online portal with data transfer capabilities. Effectiveness of the portal in improving several health outcomes from baseline-12 months will be assessed in this study.
  Interventions: Other: Electronic Patient Portal

INTERVENTIONS:
Other: Electronic Patient Portal — RelayHealth is a web-based application that allows patients and clinicians to communicate through a secure, password protected online electronic portal with data transfer capabilities. The system allows physicians and nurses to view patient questions, patient data and transmit messages to patients in response to questions or after clinic visits in an electronic message. In addition, patients can be made aware of upcoming investigations or clinic visits. Patients can also use the interface to identify any proposed changes (which would minimize recall mistakes after clinic visits) and submit queries pertaining to dialysis. Both patients and clinicians are made aware of new messages through email prompt, which moderates the asynchronous nature of electronic communication. Telephone communication can be maintained, but reserved for more urgent issues that require immediate assistance.

SUMMARY:
Home dialysis has many potential benefits compared to in-center hemodialysis including improved quality of life, reduced hospital admission and reduced cost. However, some patients perceive that home modalities are associated with increased isolation from the healthcare system, substandard care or higher risk of catastrophic events. Providing better support for home dialysis patients may enhance their ability to maintain at home, improve their health outcomes, increase quality of life and improve satisfaction with care. In other chronic disease populations a secure, online communication portal between physicians and patients has proven useful in enhancing care for patients. Thus far, the utility of an online portal communication system has not been tested in a cohort of home dialysis patients. The investigators hypothesize that this novel form of communication will improve care and outcomes for home dialysis patients. Therefore, in a cohort of home dialysis patients, the purposes of this study are as follows: 1) Does an online patient-portal improve patient satisfaction with home dialysis care? 2) Does an online patient-portal improve quality of life? 3) Does an online patient-portal reduce hospitalization and health service utilization?

DETAILED DESCRIPTION:
Home dialysis (including peritoneal dialysis and home hemodialysis) has a number of potential benefits over in-center hemodialysis (including lower healthcare costs and improved quality of life for patients). However, overall quality of life remains low compared to the general population. Furthermore, home dialysis patients (primarily those on peritoneal dialysis) continue to experience a high rate of hospitalization. Finally, there can be improvement in patient satisfaction with home dialysis, particularly in the areas of shared decision making and handling of patient requests.

Regarding satisfaction with care, peritoneal dialysis patients have identified that "attentiveness to concerns", and clarity of recommendations is important. Improved satisfaction in turn, may be associated with improvements in quality of life. Therefore, identifying novel communication systems for home dialysis patients is crucial. The use of eHealth online portals that support online communication between patients and healthcare workers is increasing. An interface that allows patients to discuss treatment plans and address clinical problems while obviating the need for telephone communication has been shown to be beneficial in some studies. Such a system may improve patient satisfaction, reduce health service utilization, and potentially improve health outcomes.

Thus far, the feasibility and potential benefit of an eHealth online portal to facilitate communication has not been evaluated in home dialysis. Therefore, in a cohort of home dialysis patients, the purpose of this study is to identify the following: 1) Does an online portal improve patient satisfaction with home dialysis care? 2) Does an online portal improve quality of life? 3) Does an online portal reduce hospitalization and health service utilization? Overall, we hope that this study will inform the need to pursue a larger, multicenter trial to more rigorously evaluate the utility of this novel form of communication for home dialysis patients.

We will conduct a prospective pilot study of prevalent (receiving home dialysis for at least three months) home dialysis patients (including both peritoneal dialysis and home hemodialysis) at Capital Health. Consecutive patients that are evaluated in the home dialysis clinic over a 4-month period will be enrolled in the study if they provide consent.

ELIGIBILITY:
Inclusion Criteria:

* Prevalent (>=3 months) home dialysis patients (peritoneal dialysis or home hemodialysis)

Exclusion Criteria:

* Does not provide consent
* On home dialysis for less than 3 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2014-10; Primary Completion 2016-02 (Actual); Study Completion 2016-02 (Actual)

PRIMARY OUTCOMES:
Change in Patient Satisfaction | 12 months
  Patient satisfaction will be examined in all patients at 0, 6 and 12 months using the Consumer Quality index (CQI) instrument (van der Veer SN, Jager KJ, Visserman E, Beekman RJ, Boeschoten EW, de Keizer NF, Heuveling L, Stronks K, Arah OA. Development and validation of the Consumer Quality index instrument to measure the experience and priority of chronic dialysis patients. Nephrol Dial Transplant. 2012 Aug;27(8):3284-91. This Dutch-language tool will be translated to English using a validated translation procedure.

SECONDARY OUTCOMES:
Change in Quality of Life | 12 Months
  Patient quality of life will be measured in all patients at 0, 6 and 12 months after initiating the study. Specifically, change from baseline in the EuroQol-5D will be evaluated at 6 and 12 months after initiation of the patient portal.
Hospitalization and Health-Care Utilization Rates | 12 Months
  Healthcare service utilization will consist of number and duration of hospitalizations, number of emergency room visits (for both dialysis and non-dialysis related complaints), number of non-advised drop-in visits to the home dialysis unit and number/duration and type of telephone contacts with the home dialysis unit. All utilization measures will be retrospectively assessed over the preceding three to twelve months (depending on available data) to get a baseline rate.

OTHER OUTCOMES:
Acceptability of Portal | 12 months
  A modified version of the Acceptability E scale (Tariman JD, Berry DL, Halpenny B, Wolpin S, Schepp K. Validation and testing of the Acceptability E-scale for web-based patient-reported outcomes in cancer care. Appl Nurs Res. 2011 Feb;24(1):53-8) will be administered at 6 and 12 months in patients utilizing the portal, to assess their perception of the tool itself.
Patient Satisfaction with the Portal | 12 months
  A secondary patient satisfaction questionnaire (Schachter ME, Bargman JM, Copland M, Hladunewich M, Tennankore KK, Levin A, Oliver M, Pauly RP, Perl J, Zimmerman D, Chan CT. Rationale for a home dialysis virtual ward: design and implementation. BMC Nephrol. 2014 Feb 14;15:33) will be used to assess patient satisfaction with the portal.

CONTACTS AND LOCATIONS:
Overall Officials: Karthik K Tennankore, MD, Principal Investigator — Capital District Health
Locations (1):
- Capital Health, Halifax, Nova Scotia, Canada

REFERENCES:
- [Derived] Kiberd J, Khan U, Stockman C, Radhakrishnan A, Phillips M, Kiberd BA, West KA, Soroka S, Chan C, Tennankore KK. Effectiveness of a Web-Based eHealth Portal for Delivery of Care to Home Dialysis Patients: A Single-Arm Pilot Study. Can J Kidney Health Dis. 2018 Sep 7;5:2054358118794415. doi: 10.1177/2054358118794415. eCollection 2018. PMID 30210802